CLINICAL TRIAL: NCT01071083
Title: Randomized Treatment Interruption of Natalizumab
Brief Title: Treatment Interruption of Natalizumab
Acronym: RESTORE
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Biogen (Industry)
Collaborators: Elan Pharmaceuticals (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 101MS205
Record Dates: First submitted 2010-02-17; First posted 2010-02-19 (Estimated); Results first posted 2013-01-30 (Estimated); Last update posted 2013-09-19 (Estimated); Status verified 2012-11

CONDITIONS: Relapsing Remitting Multiple Sclerosis
Keywords: MS
MeSH Terms: conditions — Multiple Sclerosis, Relapsing-Remitting | interventions — Natalizumab; Interferon beta-1a; Methylprednisolone; Glatiramer Acetate

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor

ARMS (3):
- natalizumab (Active Comparator)
  Interventions: Drug: natalizumab
- IV placebo (Placebo Comparator)
  Interventions: Other: IV placebo
- interferon β-1a, glatiramer acetate, or methylprednisolone (Active Comparator)
  Interventions: Drug: interferon beta 1-a; Drug: methylprednisolone; Drug: glatiramer acetate

INTERVENTIONS:
Drug: natalizumab — 300 mg intravenous every 4 weeks
  Arms: natalizumab
Drug: interferon beta 1-a — 30 ug intramuscular once per week
  Arms: interferon β-1a, glatiramer acetate, or methylprednisolone
Drug: methylprednisolone — 1000 mg intravenous every 4 weeks
  Arms: interferon β-1a, glatiramer acetate, or methylprednisolone
Other: IV placebo — placebo intravenous every 4 weeks
  Arms: IV placebo
Drug: glatiramer acetate — 20 mg subcutaneous once daily
  Arms: interferon β-1a, glatiramer acetate, or methylprednisolone

SUMMARY:
This is a randomized, rater blinded trial in patients who interrupt treatment with natalizumab with or without being treated with other immunomodulatory drugs, or continue treatment with natalizumab.

The main purpose of this study is to find out the following, when participants stop taking natalizumab for 24 weeks:

* when MS symptoms return, and
* if other drugs for MS may help control MS symptoms during the natalizumab-interruption period.

This study will also explore how quickly the effects of natalizumab return after resuming natalizumab dosing.

ELIGIBILITY:
Major criteria include:

* A diagnosis of a relapsing form of MS
* Treatment with natalizumab according to locally approved prescribing information
* Other protocol defined inclusion/exclusion criteria may apply

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 175 (Actual)
Dates: Start 2010-03; Primary Completion 2011-11 (Actual); Study Completion 2011-11 (Actual)

CONTACTS AND LOCATIONS:
Locations (30):
- United States (18):
  - Research Site, Cullman, Alabama
  - Research Site, San Francisco, California
  - Research Site, Fort Collins, Colorado
  - Research Site, Pompano Beach, Florida
  - Research Site, Atlanta, Georgia
  - Research Site, Chicago, Illinois
  - Research Site, Lake Barrington, Illinois
  - Research Site, Des Moines, Iowa
  - Research Site, Boston, Massachusetts
  - Research Site, Buffalo, New York
  - Research Site, Latham, New York
  - Research Site, Patchogue, New York
  - Research Site, Charlotte, North Carolina
  - Research Site, Raleigh, North Carolina
  - Research Site, Cleveland, Ohio
  - Research Site, Uniontown, Ohio
  - Research Site, Salt Lake City, Utah
  - Research Site, Seattle, Washington
- Germany (7):
  - Research Site, Freiburg im Breisgau, Baden-Wurttemberg
  - Research Site, München, Bavaria
  - Research Site, Hennigsdorf, Brandenburg
  - Research Site, Hamburg, Hamburg
  - Research Site, Marburg, Hesse
  - Research Site, Bochum, North Rhine-Westphalia
  - Research Site, Dresden, Saxony
- Spain (5):
  - Research Site, Barcelona, Barcelona
  - Research Site, L'Hospitalet de Llobregat, Barcelona
  - Research Site, Málaga, Malaga
  - Research Site, El Palmar, Murcia
  - Research Site, Valencia, Valencia

REFERENCES:
- [Derived] Fox RJ, Cree BAC, de Seze J, Gold R, Hartung HP, Jeffery D, Kappos L, Montalban X, Weinstock-Guttman B, Singh CM, Altincatal A, Belviso N, Avila RL, Ho PR, Su R, Engle R, Sangurdekar D, de Moor C, Fisher E, Kieseier BC, Rudick RA. Temporal Relationship Between Serum Neurofilament Light Chain and Radiologic Disease Activity in Patients With Multiple Sclerosis. Neurology. 2024 May 14;102(9):e209357. doi: 10.1212/WNL.0000000000209357. Epub 2024 Apr 22. PMID 38648580
- [Derived] Nakamura K, Brown RA, Narayanan S, Collins DL, Arnold DL; Alzheimer's Disease Neuroimaging Initiative. Diurnal fluctuations in brain volume: Statistical analyses of MRI from large populations. Neuroimage. 2015 Sep;118:126-32. doi: 10.1016/j.neuroimage.2015.05.077. Epub 2015 Jun 3. PMID 26049148

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Date of first treatment: 31 March 2010. Date of study completion: 02 November 2011.
Pre-assignment Details: 175 subjects were enrolled, all 175 were randomized.
Groups:
- Intravenous Placebo: placebo matching natalizumab, intravenous every 4 weeks
- Interferon β-1a: 30 ug intramuscular once per week
Period: Overall Study
Arm/Group | Intravenous Placebo | Natalizumab | Interferon β-1a | Glatiramer Acetate | Methylprednisolone
Started | 42 | 45 | 17 | 17 | 54
Completed | 35 | 43 | 12 | 15 | 46
Not Completed | 7 | 2 | 5 | 2 | 8
Not completed — Adverse Event | 1 | 0 | 1 | 0 | 1
Not completed — Withdrawal by Subject | 3 | 0 | 2 | 0 | 3
Not completed — Physician Decision | 1 | 0 | 0 | 1 | 1
Not completed — Early Rescue | 1 | 0 | 0 | 0 | 1
Not completed — Subject Moved | 0 | 1 | 0 | 0 | 0
Not completed — Images Not Usable (Motion) | 0 | 1 | 0 | 0 | 0
Not completed — Did Not Meet Eligibility Criteria | 0 | 0 | 1 | 1 | 1
Not completed — Did Not Want Per Protocol Treatment | 0 | 0 | 1 | 0 | 1
Not completed — Subject Refused to Continue | 1 | 0 | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Natalizumab | Intravenous Placebo | Interferon β-1a | Glatiramer Acetate | Methylprednisolone | Total
Number analyzed (Participants) | 45 | 42 | 17 | 17 | 54 | 175
Age Continuous [Mean (Standard Deviation); unit: Years] | 41.2 (9.70) | 40.0 (10.36) | 45.1 (9.92) | 44.1 (7.85) | 40.1 (9.96) | 41.2 (9.85)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 37 | 31 | 14 | 14 | 39 | 135
  Male | 8 | 11 | 3 | 3 | 15 | 40

OUTCOME MEASURES:

1. Primary Outcome: Time Course to Return of Radiological and/or Clinical Evidence of Multiple Sclerosis Activity, as Measured by the Percentage of Subjects Who Met Magnetic Resonance Imaging (MRI) and/or Clinical Relapse Rescue Criteria.
Description: Rescue criteria were: 1) central reader MRI finding of 1 new gadolinium-enhancing (Gd+) lesion of >0.8 cubic centimeters in volume or 2 or more Gd+ lesions of any size 2) clinical relapse. Clinical relapse was new or recurrent neurological symptoms not associated with fever or infection, lasting at least 24 hours, as defined by: an increase of ≥1 grade in ≥2 functional scales of the Expanded Disability Status Scale (EDSS); an increase of ≥2 grades in 1 functional scale of the EDSS; or an increase of >0.5 in EDSS if the previous EDSS was ≤5.5, or ≥0.5 if the previous EDSS was >5.5
Time Frame: 28 Weeks
Population: Of the randomized subjects, data from 167 subjects were used in efficacy analyses. Eight subjects were excluded from the analyses: 3 subjects had major protocol deviations and 5 subjects discontinued study participation prior to Week 4 Visit.
Measure: Number; unit: Percentage of subjects meeting criteria
Arm/Group | Natalizumab | Intravenous Placebo | Interferon β-1a | Glatiramer Acetate | Methylprednisolone
Number analyzed (Participants) | 45 | 41 | 14 | 15 | 52
Percentage of subjects meeting criteria | 4.7 | 60.5 | 28.6 | 53.3 | 54.8

2. Secondary Outcome: Time Course to Return of Radiological Activity, as Measured by the Percentage of Subjects Who Met Magnetic Resonance Imaging (MRI) Rescue Criteria.
Description: MRI rescue criteria were the presence of 1 new gadolinium-enhancing (Gd+) lesion of >0.8 cubic centimeters in volume or 2 or more Gd+ lesions of any size, according to the central MRI reader.
Time Frame: 28 Weeks
Population: as for outcome 1
Measure: Number; unit: Percentage of subjects meeting criteria
Arm/Group | Natalizumab | Intravenous Placebo | Interferon β-1a | Glatiramer Acetate | Methylprednisolone
Number analyzed (Participants) | 45 | 41 | 14 | 15 | 52
Percentage of subjects meeting criteria | 0.0 | 52.5 | 8.3 | 49.7 | 46.1

ADVERSE EVENTS:
Arm/Group | Intravenous Placebo | Natalizumab | Interferon β-1a | Glatiramer Acetate | Methylprednisolone
Serious Adverse Events (participants affected / at risk) | 1 | 1 | 1 | 1 | 1
Other Adverse Events (participants affected / at risk) | 35 | 38 | 15 | 15 | 42
SERIOUS ADVERSE EVENTS; cells are participants affected / at risk (number of events):
Term (organ system) | Intravenous Placebo | Natalizumab | Interferon β-1a | Glatiramer Acetate | Methylprednisolone
Chest Pain (General disorders) | 0/42 (0) | 1/45 (1) | 0/17 (0) | 0/17 (0) | 0/54 (0)
Multiple Sclerosis (Nervous system disorders) | 1/42 (1) | 0/45 (0) | 0/17 (0) | 0/17 (0) | 0/54 (0)
Multiple Sclerosis Relapse (Nervous system disorders) | 0/42 (0) | 0/45 (0) | 0/17 (0) | 1/17 (2) | 0/54 (0)
Brain Abscess (Infections and infestations) | 0/42 (0) | 0/45 (0) | 0/17 (0) | 0/17 (0) | 1/54 (1)
Syncope (Nervous system disorders) | 0/42 (0) | 0/45 (0) | 1/17 (1) | 0/17 (0) | 0/54 (0)
Presyncope (Nervous system disorders) | 0/42 (0) | 0/45 (0) | 1/17 (2) | 0/17 (0) | 0/54 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected / at risk:
Term (organ system) | Intravenous Placebo | Natalizumab | Interferon β-1a | Glatiramer Acetate | Methylprednisolone
INCISION SITE PAIN (Injury, poisoning and procedural complications) | 0/42 | 0/45 | 1/17 | 0/17 | 0/54
BACK PAIN (Musculoskeletal and connective tissue disorders) | 1/42 | 2/45 | 0/17 | 0/17 | 3/54
SYNCOPE (Nervous system disorders) | 0/42 | 0/45 | 1/17 | 0/17 | 1/54
MEMORY IMPAIRMENT (Nervous system disorders) | 2/42 | 0/45 | 1/17 | 0/17 | 0/54
FOLATE DEFICIENCY (Metabolism and nutrition disorders) | 0/42 | 0/45 | 1/17 | 0/17 | 0/54
BLOOD GLUCOSE INCREASED (Investigations) | 0/42 | 0/45 | 0/17 | 1/17 | 0/54
MUSCLE SPASMS (Musculoskeletal and connective tissue disorders) | 0/42 | 0/45 | 2/17 | 1/17 | 0/54
HYPERTENSION (Vascular disorders) | 0/42 | 0/45 | 1/17 | 0/17 | 0/54
HYPOAESTHESIA (Nervous system disorders) | 2/42 | 3/45 | 1/17 | 1/17 | 0/54
POST LUMBAR PUNCTURE SYNDROME (Injury, poisoning and procedural complications) | 1/42 | 0/45 | 2/17 | 0/17 | 2/54
DRUG SPECIFIC ANTIBODY PRESENT (Investigations) | 0/42 | 0/45 | 1/17 | 0/17 | 0/54
CONCUSSION (Injury, poisoning and procedural complications) | 0/42 | 0/45 | 0/17 | 1/17 | 0/54
HYPERREFLEXIA (Nervous system disorders) | 0/42 | 0/45 | 1/17 | 0/17 | 0/54
URINARY TRACT INFECTION (Infections and infestations) | 5/42 | 1/45 | 2/17 | 1/17 | 2/54
PROTEIN URINE PRESENT (Investigations) | 0/42 | 1/45 | 0/17 | 1/17 | 0/54
SLEEP DISORDER (Psychiatric disorders) | 0/42 | 0/45 | 1/17 | 0/17 | 3/54
DRUG HYPERSENSITIVITY (Immune system disorders) | 0/42 | 1/45 | 1/17 | 0/17 | 0/54
RASH (Skin and subcutaneous tissue disorders) | 0/42 | 1/45 | 1/17 | 0/17 | 0/54
INFLUENZA LIKE ILLNESS (General disorders) | 0/42 | 0/45 | 5/17 | 1/17 | 0/54
ECZEMA (Skin and subcutaneous tissue disorders) | 0/42 | 0/45 | 1/17 | 0/17 | 0/54
COGNITIVE DISORDER (Nervous system disorders) | 0/42 | 0/45 | 0/17 | 1/17 | 0/54
ALANINE AMINOTRANSFERASE INCREASED (Investigations) | 0/42 | 0/45 | 1/17 | 0/17 | 0/54
DYSPNOEA (Respiratory, thoracic and mediastinal disorders) | 0/42 | 0/45 | 0/17 | 1/17 | 0/54
ANTICHOLINERGIC SYNDROME (Nervous system disorders) | 0/42 | 0/45 | 0/17 | 1/17 | 0/54
BREAST CYST (Reproductive system and breast disorders) | 0/42 | 1/45 | 1/17 | 0/17 | 0/54
MULTIPLE SCLEROSIS RELAPSE (Nervous system disorders) | 8/42 | 2/45 | 4/17 | 4/17 | 11/54
HALLUCINATION, VISUAL (Psychiatric disorders) | 0/42 | 0/45 | 0/17 | 1/17 | 0/54
GAMMA-GLUTAMYLTRANSFERASE INCREASED (Investigations) | 0/42 | 0/45 | 1/17 | 0/17 | 0/54
NEURALGIA (Nervous system disorders) | 0/42 | 0/45 | 0/17 | 1/17 | 0/54
INFLUENZA (Infections and infestations) | 1/42 | 1/45 | 0/17 | 0/17 | 3/54
PANIC ATTACK (Psychiatric disorders) | 0/42 | 0/45 | 0/17 | 1/17 | 0/54
TONGUE CYST (Gastrointestinal disorders) | 0/42 | 0/45 | 1/17 | 0/17 | 0/54
SKIN LESION (Skin and subcutaneous tissue disorders) | 0/42 | 0/45 | 0/17 | 1/17 | 0/54
MUSCULAR WEAKNESS (Musculoskeletal and connective tissue disorders) | 4/42 | 2/45 | 0/17 | 0/17 | 1/54
VULVOVAGINAL CANDIDIASIS (Infections and infestations) | 0/42 | 0/45 | 0/17 | 1/17 | 0/54
CONSTIPATION (Gastrointestinal disorders) | 0/42 | 1/45 | 1/17 | 0/17 | 0/54
HYPOTENSION (Vascular disorders) | 0/42 | 0/45 | 1/17 | 0/17 | 0/54
GAIT DISTURBANCE (General disorders) | 0/42 | 0/45 | 0/17 | 1/17 | 0/54
DIZZINESS (Nervous system disorders) | 0/42 | 3/45 | 0/17 | 0/17 | 0/54
OROPHARYNGEAL PAIN (Respiratory, thoracic and mediastinal disorders) | 0/42 | 0/45 | 1/17 | 0/17 | 3/54
LACERATION (Injury, poisoning and procedural complications) | 0/42 | 0/45 | 0/17 | 1/17 | 1/54
PAIN IN EXTREMITY (Musculoskeletal and connective tissue disorders) | 1/42 | 3/45 | 0/17 | 2/17 | 1/54
INJECTION SITE HAEMATOMA (General disorders) | 0/42 | 0/45 | 0/17 | 1/17 | 0/54
UPPER RESPIRATORY TRACT INFECTION (Infections and infestations) | 6/42 | 3/45 | 0/17 | 3/17 | 6/54
WHITE BLOOD CELLS URINE POSITIVE (Investigations) | 0/42 | 0/45 | 0/17 | 1/17 | 0/54
IRON DEFICIENCY (Metabolism and nutrition disorders) | 0/42 | 0/45 | 1/17 | 0/17 | 0/54
LYMPHOCYTE MORPHOLOGY ABNORMAL (Investigations) | 0/42 | 0/45 | 0/17 | 1/17 | 0/54
NASOPHARYNGITIS (Infections and infestations) | 5/42 | 11/45 | 4/17 | 1/17 | 5/54
MIGRAINE (Nervous system disorders) | 0/42 | 0/45 | 0/17 | 1/17 | 0/54
INCREASED UPPER AIRWAY SECRETION (Respiratory, thoracic and mediastinal disorders) | 0/42 | 0/45 | 0/17 | 1/17 | 0/54
LHERMITTE'S SIGN (Nervous system disorders) | 0/42 | 0/45 | 0/17 | 1/17 | 0/54
ANXIETY (Psychiatric disorders) | 2/42 | 1/45 | 1/17 | 0/17 | 1/54
FALL (Injury, poisoning and procedural complications) | 2/42 | 1/45 | 1/17 | 1/17 | 0/54
EOSINOPHIL COUNT INCREASED (Investigations) | 0/42 | 0/45 | 1/17 | 0/17 | 0/54
BURNING FEET SYNDROME (Nervous system disorders) | 0/42 | 0/45 | 1/17 | 0/17 | 0/54
SINUS CONGESTION (Respiratory, thoracic and mediastinal disorders) | 0/42 | 0/45 | 1/17 | 0/17 | 0/54
LYMPHADENOPATHY (Blood and lymphatic system disorders) | 0/42 | 3/45 | 0/17 | 0/17 | 1/54
CONTUSION (Injury, poisoning and procedural complications) | 1/42 | 0/45 | 1/17 | 0/17 | 0/54
VITAMIN D DEFICIENCY (Metabolism and nutrition disorders) | 0/42 | 0/45 | 0/17 | 1/17 | 0/54
ARTHRALGIA (Musculoskeletal and connective tissue disorders) | 2/42 | 1/45 | 0/17 | 1/17 | 2/54
ASTHENIA (General disorders) | 0/42 | 0/45 | 2/17 | 0/17 | 0/54
HEADACHE (Nervous system disorders) | 3/42 | 8/45 | 1/17 | 1/17 | 3/54
JOINT STIFFNESS (Musculoskeletal and connective tissue disorders) | 0/42 | 0/45 | 1/17 | 1/17 | 0/54
INJECTION SITE URTICARIA (General disorders) | 0/42 | 0/45 | 0/17 | 1/17 | 0/54
DEPRESSION (Psychiatric disorders) | 2/42 | 1/45 | 1/17 | 0/17 | 0/54
FATIGUE (General disorders) | 6/42 | 2/45 | 1/17 | 2/17 | 2/54
INJECTION SITE PAIN (General disorders) | 0/42 | 0/45 | 0/17 | 1/17 | 0/54
PRESYNCOPE (Nervous system disorders) | 0/42 | 0/45 | 1/17 | 0/17 | 0/54
FUNGAL SKIN INFECTION (Infections and infestations) | 0/42 | 0/45 | 1/17 | 0/17 | 0/54
DYSGEUSIA (Nervous system disorders) | 0/42 | 0/45 | 1/17 | 0/17 | 0/54
PARAESTHESIA (Nervous system disorders) | 3/42 | 3/45 | 0/17 | 0/17 | 0/54
DEHYDRATION (Metabolism and nutrition disorders) | 0/42 | 1/45 | 0/17 | 1/17 | 0/54
PYELONEPHRITIS (Infections and infestations) | 0/42 | 0/45 | 0/17 | 1/17 | 0/54
BALANCE DISORDER (Nervous system disorders) | 1/42 | 0/45 | 0/17 | 1/17 | 0/54
PRODUCTIVE COUGH (Respiratory, thoracic and mediastinal disorders) | 0/42 | 0/45 | 1/17 | 0/17 | 0/54
NAUSEA (Gastrointestinal disorders) | 0/42 | 1/45 | 1/17 | 0/17 | 0/54

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The provisions of our agreement are subject to confidentiality but generally the PI can publish, for noncommercial purposes only, results and methods of the trial, but no other Sponsor Confidential Information. PI must give Sponsor no less than 60 days to review any manuscript for a proposed publication and must delay publication for up to 90 days thereafter if Sponsor needs to file any patent application to protect any of Sponsor's intellectual property contained in the proposed publication.